CLINICAL TRIAL: NCT01097486
Title: Phase 2 Study Evaluating Safety and Preliminary Efficacy of NeoFuse When Combined With MasterGraft Matrix in Subjects Undergoing Multi-Level Anterior Cervical Discectomy and Fusion With Anterior Cervical Plate Fixation
Brief Title: Safety and Preliminary Efficacy Study of NeoFuse in Subjects Undergoing Multi-Level Anterior Cervical Discectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mesoblast, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MSB-CF002
Record Dates: First submitted 2010-03-30; First posted 2010-04-01 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2016-12

CONDITIONS: Cervical Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis
Keywords: Cervical Degenerative Disc Disease; Degenerative Spondylolisthesis; Spinal Stenosis; Stem cells; Adult Stem Cells; Anterior cervical discectomy and Fusion (ACDF); Cervical Allograft Spacer; Anterior Cervical Plate Fixation
MeSH Terms: conditions — Spinal Stenosis | interventions — Gene Fusion; Transplantation, Homologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allograft (Active Comparator): Cervical Spinal Fusion with Allograft
  Interventions: Procedure: Allograft
- NeoFuse (Experimental): Cervical Spinal Fusion with NeoFuse
  Interventions: Biological: NeoFuse

INTERVENTIONS:
Biological: NeoFuse — Single Dose NeoFuse Surgical Implantation
  Other Names: Anterior Cervical Discectomy and Fusion with NeoFuse; Cervical Spinal Fusion; Stem Cells
  Arms: NeoFuse
Procedure: Allograft — Single Dose Allograft Surgical Implantation
  Other Names: Anterior Cervical Discectomy and Fusion with Allograft; Cervical Spinal Fusion; Control
  Arms: Allograft

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of NeoFuse in subjects with a diagnosis of degenerative disc disease (DDD) at 2 or more adjacent cervical vertebral levels between C3-C4 to C7-T1. All subjects in this study will undergo 2 or 3 level anterior cervical discectomy and fusion with anterior cervical plate fixation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, single-blinded, controlled study evaluating safety and preliminary efficacy of immunoselected, culture-expanded, nucleated, allogeneic MPCs (NeoFuse) combined with MasterGraft Matrix in a commercially available PEEK cervical spacer compared to a cervical Allograft Spacer control in subjects undergoing 2 or 3 level anterior cervical discectomy and fusion with anterior cervical plate fixation.

After the screening and surgical visits, each subject will be evaluated clinically and radiographically within 3 days and 30 days after surgery, and at 3, 6, 12, and 24 months after surgery.

Subjects will be evaluated at the same time points for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females between 18 and 70 years of age, inclusive.
2. Has the ability to understand the requirements of the study, to provide written informed consent, and to comply with the study protocol.
3. Has the ability to understand and provide written authorization for the use and disclosure of personal health information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) privacy ruling in the US].
4. Has a documented symptomatic diagnosis of DDD at C3-C4 to C7-T1.
5. Has symptomatic radiculopathy and/or myelopathy correlating to radiographic findings of duration of 6 weeks or greater that had failed to respond to non-operative management
6. Is a candidate for anterior cervical discectomy and fusion in two or three adjacent cervical interbody levels between C3-C4 to C7-T1
7. Has a stable screening electrocardiogram (ECG), as determined by the investigator that would not preclude surgery.

Exclusion Criteria:

1. Female subjects who are pregnant or nursing, or women planning to become pregnant during the first year (12 months) following surgery.
2. Has a current or prior history within the last 3 years of neoplasm (excluding basal cell carcinoma) and/or any active neoplasm within the last 24 months, prior to screening.
3. Has at the time of surgery a systemic or local infection at the site of proposed surgery.
4. Has or is undergoing revision of a prior fusion surgery at any involved level.
5. Requires ACDF at only one cervical interbody level or more than 3 adjacent cervical interbody levels.
6. Requires ACDF without the use of an anterior cervical plating system.
7. Has osteoporosis as defined by a DEXA T score of ≤ -3.0 or a history of fragility fractures or other significant bone disease contraindicating the use of spinal instrumentation.
8. Has a documented medical history or radiographic evidence of a metabolic bone disease or other condition which would negatively impact the bone healing process.
9. Has a positive screen for human immunodeficiency virus (HIV) antibodies.
10. has had treatment with any investigational therapy or device within 6 months of study surgery and/or plans to participate in any other allogeneic stem cell/progenitor cell therapy trial during the 2-year follow-up period.
11. Has been a recipient of prior stem cell/progenitor cell therapy for spinal fusion surgery.
12. Has 20% or greater anti-human leukocyte antigen (HLA) antibody titer and/or has antibody specificities to donor HLA antigens.
13. Is transient or has been treated in the last 6 months before enrollment for alcohol and/or drug abuse in an inpatient substance abuse program.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety of NeoFuse using physical examinations, vital signs, treatment emergent adverse events (TEAEs), and the results of clinical lab tests (hematology, serum chemistry, inflammation, and and immunology). | 2 years

SECONDARY OUTCOMES:
To evaluate the fusion success with NeoFuse compared to allograft spacer using CT scans and x-ray of the involved cervical spine levels and assess the change in outcomes (NDI, SF-36, Zung Depression Questionnaire, and WPAI. | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Brown, Study Director — Mesoblast, Ltd.
Locations (8):
- United States (8):
  - UC Davis Spine Center, Sacramento, California
  - The Spine Institute, Santa Monica, California
  - Denver Spine, Denver, Colorado
  - Rocky Mountain Associates in Orthopedic Medicine, P.C., Loveland, Colorado
  - Tallahassee Neurological Clinic, P.A., Tallahassee, Florida
  - Fort Wayne Orthopaedics, Fort Wayne, Indiana
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - Central Texas Spine Institute, Austin, Texas

REFERENCES:
- See also: Sponsor Website — http://www.mesoblast.com